CLINICAL TRIAL: NCT05253716
Title: The Effects of Immunonutritional Supplement After Total Gastrectomy in Patients With Stage III Gastric Cancer on Long-term Disease-free Survival After Total Gastrectomy in Patients With Stage III Gastric Cancer
Brief Title: Immunonutritional Supplement After Total Gastrectomy in Patients With Stage III Gastric Cancer
Acronym: CRUCIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated cancer hospital of Nanjing Medical University (Unknown); Nanjing Jiangning Hospital (Unknown); Zhenjiang First People's Hospital (Other); The Third Affiliated Hospital of Soochow University (Other); ChangZhou Second hospital (Unknown); The First Affiliated Hospital of Soochow University (Other); Second Affiliated Hospital of Soochow University (Other); Yixing People's Hospital (Other); The Second Hospital of Nanjing Medical University (Other); Wuxi People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Xinying, Prof., Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12-4
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Stage III Gastric Cancer
Keywords: Oral nutritional supplement; Immunonutrition; long-term survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immune nutrition support (Experimental): In the immune nutrition support group, in addition to diet, and patients will also consume two bottles per day of a high-calorie, high-protein ONS and three capsules of fish oil after discharge lasted for 6 months.
  Interventions: Other: ONS
- control (No Intervention): In the control group, patients will receive nutrition counseling in addition to diet.

INTERVENTIONS:
Other: ONS — Immunonutritional supplement
  Other Names: fish oil
  Arms: immune nutrition support

SUMMARY:
Gastric cancer patients with stage III will be randomized to immune nutrition support or control group at discharge after total gastrectomy. Patients will receive 6 months of immune nutrition support or normal diet after discharge. The primary and secondary outcomes will be collected.

DETAILED DESCRIPTION:
Gastric cancer patients with stage III after total gastrectomy at discharge, if she/he has nutrition risk (NRS2002≥3), then she/he will be randomized to immune nutrition support (INS) or control (C) group after discharge. In the INS group, in addition to diet, and patients will also consume two bottles per day of a high-calorie, high-protein ONS and three capsules of fish oil lasted for 6 months. In the C group, patients will receive normal diet. Both groups will receive nutrition counseling.

The primary and secondary outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of patients or their legal representatives to participate in this study
2. consecutive adult (≥18 years) patients underwent radical gastrectomy (total gastrectomy) with pathological TNM stage III
3. nutrition Risk Screening (NRS) 2002≥3 at discharge
4. eastern Cooperative Oncology Group (ECOG) score of 0-2 at discharge

Exclusion Criteria:

1. unable to oral or consume ONS
2. has received neoadjuvant chemotherapy
3. pregnancy
4. palliative surgery or gastric stump cancer or Borrmann type IV
5. oral anticoagulants cannot be stopped; congenital acquired immune deficiency disease
6. serious cardiovascular disease including chronic heart failure, angina pectoris, myocardial infarction, arrhythmias (such as atrial fibrillation), or uncontrolled hypertension
7. severe liver and kidney diseases including active hepatitis, cirrhosis, and uremia
8. diabetes has developed complications or uncontrolled by medications
9. previous use of drugs affecting immune function
10. previous use of fish oil capsule > 2 times / week or contraindications to fish oil capsule
11. motor system diseases cannot complete grip strength measurement and 5-time chair stand test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival after discharge | up to 3 years
  from date of randomization to disease recurrence or death

SECONDARY OUTCOMES:
3-year overall survival | up to 3 years.
  from date of randomization to death due to any reason,
unplanned readmission rate | up to 6 months.
  readmission due to unplanned reason
Quality of life after discharge | up to 12 months.
  Quality of life assessed by EORTC QLQ-C30
incidence of sarcopenia after discharge | up to 12 months.
  sarcopenia is defined as low skeletal muscle mass plus low muscle strength or low physical ability.
Changes in BMI (weight and height will be combined to report BMI in kg/m^2) | up to 12 months.
  nutritional status after discharge
Changes in albumin level | up to 12 months.
  nutritional status after discharge
Changes in prealbumin level | up to 12 months.
  nutritional status after discharge
Changes in hemoglobin level | up to 12 months.
  nutritional status after discharge
Changes in weight | up to 12 months.
  nutritional status after discharge
toxicity of chemotherapy graded according to the CTCAE, version 5.0 | up to 6 months.
  Chemotherapy toxicity will be monitored at end of each cycle during chemotherapy by investigators, and graded according to the CTCAE, version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, MD, Principal Investigator — Jinling Hosptial
Locations (1):
- Jinling Hospital, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heneghan HM, Zaborowski A, Fanning M, McHugh A, Doyle S, Moore J, Ravi N, Reynolds JV. Prospective Study of Malabsorption and Malnutrition After Esophageal and Gastric Cancer Surgery. Ann Surg. 2015 Nov;262(5):803-7; discussion 807-8. doi: 10.1097/SLA.0000000000001445. PMID 26583669
- [Background] Huang DD, Cai HY, Chen XY, Dong WX, Wangchuk D, Yan JY, Chen XL, Dong QT. Value of Sarcopenia defined by the new EWGSOP2 consensus for the prediction of Postoperative Complications and Long-term Survival after Radical Gastrectomy for Gastric Cancer: A comparison with four common nutritional screening tools. J Cancer. 2020 Aug 6;11(19):5852-5860. doi: 10.7150/jca.49815. eCollection 2020. PMID 32913478
- [Background] Zheng HL, Lu J, Li P, Xie JW, Wang JB, Lin JX, Chen QY, Cao LL, Lin M, Tu R, Huang CM, Zheng CH. Effects of Preoperative Malnutrition on Short- and Long-Term Outcomes of Patients with Gastric Cancer: Can We Do Better? Ann Surg Oncol. 2017 Oct;24(11):3376-3385. doi: 10.1245/s10434-017-5998-9. Epub 2017 Jul 11. PMID 28699132
- [Background] Ongaro E, Buoro V, Cinausero M, Caccialanza R, Turri A, Fanotto V, Basile D, Vitale MG, Ermacora P, Cardellino GG, Nicoletti L, Fornaro L, Casadei-Gardini A, Aprile G. Sarcopenia in gastric cancer: when the loss costs too much. Gastric Cancer. 2017 Jul;20(4):563-572. doi: 10.1007/s10120-017-0722-9. Epub 2017 May 5. PMID 28477106
- [Background] Park JH, Kim E, Seol EM, Kong SH, Park DJ, Yang HK, Choi JH, Park SH, Choe HN, Kweon M, Park J, Choi Y, Lee HJ. Prediction Model for Screening Patients at Risk of Malnutrition After Gastric Cancer Surgery. Ann Surg Oncol. 2021 Aug;28(8):4471-4481. doi: 10.1245/s10434-020-09559-3. Epub 2021 Jan 22. PMID 33481124
- [Background] Oh SE, Choi MG, Seo JM, An JY, Lee JH, Sohn TS, Bae JM, Kim S. Prognostic significance of perioperative nutritional parameters in patients with gastric cancer. Clin Nutr. 2019 Apr;38(2):870-876. doi: 10.1016/j.clnu.2018.02.015. Epub 2018 Feb 20. PMID 29503057
- [Background] Lee JK, Park YS, Lee K, Youn SI, Won Y, Min SH, Ahn SH, Park DJ, Kim HH. Prognostic significance of surgery-induced sarcopenia in the survival of gastric cancer patients: a sex-specific analysis. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1897-1907. doi: 10.1002/jcsm.12793. Epub 2021 Sep 17. PMID 34533290
- [Background] Muscaritoli M, Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Oldervoll L, Ravasco P, Solheim TS, Strasser F, de van der Schueren M, Preiser JC, Bischoff SC. ESPEN practical guideline: Clinical Nutrition in cancer. Clin Nutr. 2021 May;40(5):2898-2913. doi: 10.1016/j.clnu.2021.02.005. Epub 2021 Mar 15. PMID 33946039
- [Background] Miyazaki Y, Omori T, Fujitani K, Fujita J, Kawabata R, Imamura H, Okada K, Moon JH, Hirao M, Matsuyama J, Saito T, Takahashi T, Kurokawa Y, Yamasaki M, Takiguchi S, Mori M, Doki Y; Osaka University Clinical Research Group for Gastroenterological Study. Oral nutritional supplements versus a regular diet alone for body weight loss after gastrectomy: a phase 3, multicenter, open-label randomized controlled trial. Gastric Cancer. 2021 Sep;24(5):1150-1159. doi: 10.1007/s10120-021-01188-3. Epub 2021 Apr 9. PMID 33835329
- [Background] Meng Q, Tan S, Jiang Y, Han J, Xi Q, Zhuang Q, Wu G. Post-discharge oral nutritional supplements with dietary advice in patients at nutritional risk after surgery for gastric cancer: A randomized clinical trial. Clin Nutr. 2021 Jan;40(1):40-46. doi: 10.1016/j.clnu.2020.04.043. Epub 2020 Jun 2. PMID 32563598
- [Background] Huang YH, Chiu WC, Hsu YP, Lo YL, Wang YH. Effects of Omega-3 Fatty Acids on Muscle Mass, Muscle Strength and Muscle Performance among the Elderly: A Meta-Analysis. Nutrients. 2020 Dec 4;12(12):3739. doi: 10.3390/nu12123739. PMID 33291698
- [Background] Ortega L, Lobos-Gonzalez L, Reyna-Jeldes M, Cerda D, De la Fuente-Ortega E, Castro P, Bernal G, Coddou C. The Omega-3 fatty acid docosahexaenoic acid selectively induces apoptosis in tumor-derived cells and suppress tumor growth in gastric cancer. Eur J Pharmacol. 2021 Apr 5;896:173910. doi: 10.1016/j.ejphar.2021.173910. Epub 2021 Jan 26. PMID 33508285
- [Background] Lu Z, Fang Y, Liu C, Zhang X, Xin X, He Y, Cao Y, Jiao X, Sun T, Pang Y, Wang Y, Zhou J, Qi C, Gong J, Wang X, Li J, Tang L, Shen L. Early Interdisciplinary Supportive Care in Patients With Previously Untreated Metastatic Esophagogastric Cancer: A Phase III Randomized Controlled Trial. J Clin Oncol. 2021 Mar 1;39(7):748-756. doi: 10.1200/JCO.20.01254. Epub 2021 Jan 8. PMID 33417481
- [Derived] Zhou D, Liu Y, Zhang L, Lu M, Gao X, Li G, Xiang X, Xu H, Li G, Sun Z, Wei W, Yi K, Zuo J, Wu Y, Qian J, Zhou J, Duan K, Wu Y, Tian Z, Jiang C, Wang X. Effects of oral immunonutritional supplement on 3-year disease-free survival in gastric cancer patients with pathological stage III after total gastrectomy (CRUCIAL): study protocol of a multicentre, randomised clinical trial. BMJ Open. 2023 Apr 11;13(4):e067990. doi: 10.1136/bmjopen-2022-067990. PMID 37041057